CLINICAL TRIAL: NCT01264926
Title: Evaluation of the Difference in the Acromion Humerus Gap at Sitting,Lying
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: saf004-CTIL-HMO
Record Dates: First submitted 2010-12-16; First posted 2010-12-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Shoulder Impingement Syndrome.
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rotator cuff tear, pain

SUMMARY:
The Objective is to evaluation the difference between the upper end of the Humerus head and the bottom end of the Acromion in sitting and lying, and to examine this difference to shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* men and women with or without shoulder pain.

Exclusion Criteria:

* unwillingness to sign informed consent

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: men and women with or without shoulder pain0
Sampling Method: Non-Probability Sample
Dates: Start 2012-02; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
level of pain as measured by the visual analogue score